CLINICAL TRIAL: NCT06727357
Title: Clinical Utility of a Next Generation Sequencing-based "Oncochip" for Therapeutic Decision in Metastatic Breast Cancer. Study SHARP
Brief Title: Next Generation Sequencing-based "Oncochip" for Therapeutic Decision in Metastatic Breast Cancer. Study SHARP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IEO 674
Record Dates: First submitted 2024-11-21; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer, Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AZD2014 (Experimental): Selective and potent inhibitor of mTOR kinase
  Interventions: Drug: Chemotherapy
- Selumetinib (Experimental): selective and potent inhibitor of MEK1/2 kinases
  Interventions: Drug: Chemotherapy
- Olaparib (Experimental): Inhibitor of the PARP enzyme involved in DNA repair
  Interventions: Drug: Chemotherapy
- Bicalutamide (Experimental): nonsteroidal antiandrogen
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — in according to institutional guidelines

SUMMARY:
The present trial clinical proposes to randomize patients with cancer metastatic disease of the breast progressing on standard therapy to receive a treatment selected from 4 "targeted" drugs (a MEK kinase inhibitor, an mTOR kinase inhibitor, an of the enzyme involved in DNA repair PARP and an androgen receptor inhibitor) on the basis of possible presence of mutations in a panel of 61 genes analyzed on metastatic tissue from biopsy, or receive standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients (women or men) with histologically confirmed metastatic breast cancer
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Written informed consent obtained prior to enrollment
* Age ≥ 18 years
* Blood and tumor tissue sample available for research
* Measurable disease
* Other site accessible for biopsy, except bone lesions if this is the only accessible site, or biopsy obtained within the previous 6 months
* Medical history, blood parameters and clinical conditions do not indicate major dysfunctions of organ

To treatment:

- Maintenance of screening inclusion criteria

Exclusion Criteria:

* Presence of visceral crisis, defined according to ABC3/ESMO guidelines
* Patients with local recurrence that can be treated with surgery and/or radiotherapy alone
* Patients who have previously received palliative radiotherapy on the only site accessible to biopsy
* Patients with metastatic disease limited to bone
* Patients with metastatic disease limited to the brain, unless planned a surgical excision, in which case tissue can be collected for screening
* Severe hematopoietic, renal and/or hepatic insufficiency
* Known contraindication to biopsy
* Neoplastic pathology of different histology in the previous 5 years, except carcinoma in situ of cervical basal or squamous cell carcinoma of the skin, if adequately treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Comparison of progression-free survival | from baseline to the end of treatment (up to 12 months)
  Comparison of progression-free survival in the experimental arm vs control arm

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Curigliano, MD, Principal Investigator — Istituto Eur
Locations (1):
- Istituto Europeo di Oncologia, Milan, Italy